CLINICAL TRIAL: NCT03821649
Title: Protocol for a Mixed Methods Feasibility Study for the Surviving Opioid Overdose With Naloxone Education and Resuscitation (SOONER) Trial
Brief Title: SOONER Feasibility Study Protocol
Acronym: SOONER
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Unity Health Toronto (Other)
Collaborators: OCAD University (Other); Toronto Public Health (Other Government)
Responsible Party: Sponsor
Allocation: Randomized | Model: Single Group | Masking: Single | Purpose: Other
Other Study IDs: 1
Record Dates: First submitted 2019-01-17; First posted 2019-01-30 (Actual); Last update posted 2022-05-23 (Actual); Status verified 2022-05

CONDITIONS: Overdose
Keywords: Education; Naloxone; Opioid; Overdose; Resuscitation
MeSH Terms: conditions — Drug Overdose | interventions — Residence Characteristics

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- SOONER Training and Naloxone Kit (Experimental): Participants in this arm will be shown the SOONER overdose response training video at the time of recruitment and given the SOONER Naloxone kit to take home.
  Interventions: Behavioral: SOONER Training and Naloxone Kit Kit
- Community or Hospital-Based Training (Active Comparator): Control arm - participants in this arm will be referred to the standard of care for Naloxone training. This standard of care includes community-based OEND programs and/or an existing hospital-based OEND program..
  Interventions: Behavioral: Community or Hospital-Based Training

INTERVENTIONS:
Behavioral: SOONER Training and Naloxone Kit Kit — Participants are shown our unique overdose response education video and given the associated kit to take home.
  Arms: SOONER Training and Naloxone Kit
Behavioral: Community or Hospital-Based Training — Referral to standard of care for Naloxone training
  Arms: Community or Hospital-Based Training

SUMMARY:
Opioid Overdose Education and Naloxone Distribution programs (OEND) involve training and equipping people who are likely to be bystanders to opioid overdose to recognize and respond to opioid-related emergencies by activating emergency services, delivering basic life support and administering naloxone. The goal of the Surviving Opioid Overdose with Naloxone Education and Resuscitation (SOONER) trial is to identify if point-of-care OEND increases rates of satisfactory bystander resuscitative performance to simulated opioid overdose in comparison with the existing standard of care. Recruitment and retention of participants at risk of overdose, and the acceptability of the simulated overdose outcome may challenge the feasibility of the SOONER trial. The primary objective is to identify if an integrated participant recruitment and retention strategy can recruit approximately 28 eligible participants within 4 weeks and maintain less than 50% attrition in the context of a randomized trial on point-of-care OEND and simulated overdose resuscitation performance in family practice, emergency department, and addictions settings in Toronto, Ontario. After the initial 28 participants, we are continuing to recruit up to 50 more participants in a bridging phase that leads into the full trial.

DETAILED DESCRIPTION:
Deaths from opioid overdose represent an important and expanding global public health epidemic. Opioid Overdose Education and Naloxone Distribution programs (OEND) involve training and equipping people who are likely to witness overdose to recognize these emergencies and administer essential first aid interventions including naloxone, a widely known and effective competitive opioid antagonist. Policymakers and practitioners have called for expanded access to OEND programs in clinical settings such as emergency departments, family practice, and addiction medicine clinics, or "point-of-care OEND". Point-of-care OEND would improve access to this potentially life-saving intervention. Simple and effective point-of-care OEND tools are a prerequisite for the successful translation of this intervention into general ambulatory settings, including family practice, addiction medicine and psychiatry clinics, and emergency departments. The investigators plan to conduct a randomized trial to evaluate the educational effectiveness of a novel point-of-care OEND kit in a simulated opioid overdose, in comparison with existing community- and hospital-based OEND programs.

Conducting trials among people who use drugs or who are likely to witness overdose involves several well-documented scientific, logistical, and bioethical challenges. These challenges contribute to the persistent under-evaluation of interventions to enhance the health of this marginalized population, and threats to study validity when retention rates are low.

Recruitment, retention and attrition rates could alter the study timelines, logistics and costs for the proposed trial. A feasibility study is needed to evaluate and refine an integrated participant recruitment and retention strategy, develop expected retention rates, establish the local acceptability of study procedures in recruitment sites, and reconsider study design and analysis if required. A feasibility study will also permit the evaluation of basic randomization and data collection procedures.

The primary objective of this feasibility study is to identify if an integrated participant recruitment and retention strategy can recruit approximately 28 eligible participants within 4 weeks and maintain less than 50% attrition in the context of a randomized trial on point-of-care OEND and simulated overdose resuscitation performance in family practice, emergency department, and addiction medicine settings at St. Michael's Hospital, and in family practice at the Inner City Family Health Team.

ELIGIBILITY:
Participants are eligible by meeting any one or more of the following:

1. Have a history of taking opioids at recognized 'high doses' (whether by prescription or otherwise, defined as >100mg morphine equivalent per day).
2. Live with or is in frequent contact with others who use opioids or heroin.
3. Have required emergency care for opioid overdose previously.
4. Are enrolled in opioid agonist treatment programs (or has been in the last 6 months), including methadone or buprenorphine maintenance programs, particularly at high risk periods such as induction or discharge.
5. Are being released from prison, and have a history of non-medical opioid use.
6. Are receiving prescription opioid therapy with risk factors for adverse effects, including relevant comorbidities, co-prescriptions of benzodiazepines or other sedatives, concomitant ongoing alcohol use, or high dose prescription opioid therapy.
7. Uses non-medical opioids, injects opioids, or acquires opioids from sources other than a pharmacy or healthcare setting.

Exclusion Criteria: Participants are ineligible by meeting any one or more of the following:

1. Have a community do not resuscitate order.
2. Have a terminal illness, end-of-life care, or illness likely to result in death within the study period.
3. Have no mode of contact or follow-up.
4. Plan to move away from Toronto during the study period.
5. Have insufficient English language skills to participate in the study.
6. Are an active or previously practicing healthcare professional or professional first responder (e.g.: firefighter, police officer, lifeguard, industrial first responder).

Min Age: 16 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 90 (Actual)
Dates: Start 2019-01-23 (Actual); Primary Completion 2020-03-01 (Actual); Study Completion 2020-12-10 (Actual)

PRIMARY OUTCOMES:
Participant recruitment rate (participants recruited in 4 weeks) | 4 weeks
  Approximately 28 participants are recruited within 4 weeks.
  The recruitment and retention strategy will be deemed "feasible" if BOTH of the following conditions are met:
  (A) approximately 28 participants are recruited within 4 weeks, AND (B) there is less than 50% attrition at the underlying study's outcome simulation.
Participant attrition at the underlying study's outcome simulation | 4-6 weeks
  less than 50% attrition at the underlying study's outcome simulation.
  Primary outcome description: The recruitment and retention strategy will be deemed "feasible" if BOTH of the following conditions are met:
  (A) approximately 28 participants are recruited within 4 weeks, AND (B) there is less than 50% attrition at the underlying study's outcome simulation.

SECONDARY OUTCOMES:
Site recruitment rates | 28 days
  Rate of participant recruitment in each of the family practice, emergency department, and addiction medicine sites associated with a single academic health care centre.
Participant retention rates | 4-6 weeks
  Comparison of retention rate between intervention and control arms
Descriptions of study process problems | 4-6 weeks
  Semi-structured interviews with study participants and unstructured verbal and written feedback from study and recruitment site staff concerning challenges and opportunities for improving any study processes (including participant recruitment, randomization, implementation of the intervention and control, retention, follow-up, outcome assessment and data collection).

CONTACTS AND LOCATIONS:
Locations (4):
- Canada (4):
  - Inner City Family Health Team, Toronto, Ontario
  - St Michael's Hospital Emergency Department, Toronto, Ontario
  - St Micheal's Health Centre at 410, Toronto, Ontario
  - St Micheal's Hospital Rapid Access Addictions Medicine Clinic, Toronto

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] United Nations Office on Drugs and Crime, World Health Organization. Discussion paper UNODC/WHO 2013: Opioid overdose: preventing and reducing opioid overdose mortality. 2013; Available at: http://www.unodc.org/docs/treatment/overdose.pdf. Accessed 04/23, 2014. Archived by WebCite© at http://www.webcitation.org/6U3qbjl2E)
- [Background] Clark AK, Wilder CM, Winstanley EL. A systematic review of community opioid overdose prevention and naloxone distribution programs. J Addict Med. 2014 May-Jun;8(3):153-63. doi: 10.1097/ADM.0000000000000034. PMID 24874759
- [Background] Doyon S, Aks SE, Schaeffer S. Expanding access to naloxone in the United States. J Med Toxicol. 2014 Dec;10(4):431-4. doi: 10.1007/s13181-014-0432-1. No abstract available. PMID 25316516
- [Background] Beletsky L, Ruthazer R, Macalino GE, Rich JD, Tan L, Burris S. Physicians' knowledge of and willingness to prescribe naloxone to reverse accidental opiate overdose: challenges and opportunities. J Urban Health. 2007 Jan;84(1):126-36. doi: 10.1007/s11524-006-9120-z. PMID 17146712
- [Background] Coffin PO, Fuller C, Vadnai L, Blaney S, Galea S, Vlahov D. Preliminary evidence of health care provider support for naloxone prescription as overdose fatality prevention strategy in New York City. J Urban Health. 2003 Jun;80(2):288-90. doi: 10.1093/jurban/jtg031. PMID 12791804
- [Background] Meyers K, Webb A, Frantz J, Randall M. What does it take to retain substance-abusing adolescents in research protocols? Delineation of effort required, strategies undertaken, costs incurred, and 6-month post-treatment differences by retention difficulty. Drug Alcohol Depend. 2003 Jan 24;69(1):73-85. doi: 10.1016/s0376-8716(02)00252-1. PMID 12536068
- [Derived] Parsons JA, Markowitz B, Thomas R, Norris K, Charles M, King C, Sellen K, Campbell DM, Leece P, Klaiman M, Chapman L, Hopkins S, Shahin R, Handford C, Stergiopoulos V, Morrison LJ, Strike C, Orkin AM; SOONER investigators. The opportunity to save a life: A qualitative study of a point-of-care overdose education and naloxone distribution intervention. PLoS One. 2025 Jun 25;20(6):e0326495. doi: 10.1371/journal.pone.0326495. eCollection 2025. PMID 40560908
- [Derived] Orkin AM, Charles M, Norris K, Thomas R, Chapman L, Wright A, Campbell DM, Handford C, Klaiman M, Hopkins S, Shahin R, Thorpe K, Juni P, Parsons J, Sellen K, Goso N, Hunt R, Leece P, Morrison LJ, Stergiopoulos V, Turner S, Strike C. Mixed methods feasibility study for the surviving opioid overdose with naloxone education and resuscitation (SOONER) trial. Resusc Plus. 2021 May 14;6:100131. doi: 10.1016/j.resplu.2021.100131. eCollection 2021 Jun. PMID 34223388
- [Derived] Orkin A, Campbell D, Handford C, Hopkins S, Klaiman M, Leece P, Parsons JA, Shahin R, Strike C, Thorpe K, Sellen K, Milos G, Wright A, Charles M, Sniderman R, Morrison L; SOONER Investigators. Protocol for a mixed-methods feasibility study for the surviving opioid overdose with naloxone education and resuscitation (SOONER) randomised control trial. BMJ Open. 2019 Nov 12;9(11):e029436. doi: 10.1136/bmjopen-2019-029436. PMID 31722937